CLINICAL TRIAL: NCT01536678
Title: Bioequivalence of Two Levothyroxine Tablet Formulations in Healthy Indian Volunteers: A Single-dose, Randomized, Open-label, Crossover Study
Brief Title: Bioequivalence of Two Levothyroxine Tablet Formulations in Healthy Indian Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 116526
Record Dates: First submitted 2012-02-02; First posted 2012-02-22 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2012-10

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test formulation of levothyroxine (Active Comparator): Single dose of 600 mcg of levothyroxine administered in dosing period 1 or 2..
  Interventions: Drug: Levothyroxine
- Reference formulation of levothyroxine (Active Comparator): Single dose of 600 mcg of levothyroxine administered in dosing period 1 or 2.
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine — Single dose of 600mcg of test formulation of levothyroxine administered in dosing period 1 or 2.
  Arms: Test formulation of levothyroxine
Drug: Levothyroxine — Single dose of 600mcg of reference formulation of levothyroxine administered in dosing period 1 or 2.
  Arms: Reference formulation of levothyroxine

SUMMARY:
GSK markets a drug called levothyroxine or T4 that is used to treat patients with hypothyroidism. Till date, the active drug substance or active pharmaceutical ingredient (API) for levothyroxine tablets marketed in India has been obtained from a particular source. GSK India proposes to change the source of the API from the existing source to a new source. Some patients may experience a change in clinical effect when switched from one formulation to another. Therefore this study is being done to understand whether a change in API in levothyroxine tablet has any impact on the clinical effect of the drug.

The purpose of this study is to:

See how quickly the levothyroxine tablet from the new source (single dose of 600mcg) enters the bloodstream, is distributed in the body, broken down and removed compared to the levothyroxine tablet from the existing source (single dose of 600mcg).

Study the effect of single 600mcg doses of levothyroxine tablet from new source and levothyroxine tablet from existing source on TSH level in the blood.

Study the safety and side effects of single 600mcg doses of levothyroxine tablet from new source and levothyroxine tablet from existing source.

DETAILED DESCRIPTION:
Levothyroxine (T4) is used to treat patients with hypothyroidism and may often result in lifelong therapy. Its physiologically active metabolite is tri-iodothyronine (T3). Levothyroxine is also endogenously produced in the body. Since small changes in levothyroxine administration (e.g. change in brand or formulation) can cause significant changes in serum thyroid stimulating hormone (TSH) concentrations, precise and accurate TSH control is critical to avoid potential adverse iatrogenic effects. Till date, the active pharmaceutical ingredient (API) for levothyroxine tablets marketed in India has been sourced from company 1. GSK India proposes to change the source of the API from the existing source (company 1) to to new source (company 2). In view of this change in the source of API, it is essential to determine whether it has any impact on drug product performance based on pharmacokinetic (PK) measures of total serum T4 and total serum T3 of the to-be-marketed formulation of levothyroxine (test formulation from company 2, Treatment A) relative to the formulation currently in the market (reference formulation from company 1, Treatment B).

This will be a single-center, open-label, two-period, two-treatment, two-sequence, randomized, single-dose, crossover study. 26 healthy adult males will be randomized to receive a single dose (6 x 100mcg tablets = 600mcg) of the test formulation of levothyroxine and reference formulation of levothyroxine separately in each treatment period. There will be two treatment sequences (AB, BA) and a 35 day washout between the two treatment periods.

The study will be conducted at BA/BE facility after approval from an independent ethics committee. Subjects will have a screening visit within 21 days prior to the first dose of study drug, two treatment periods with each containing a single dose of study drug, followed by 48 hours of serial PK sample collection. Subjects will check out of the unit on Day 3 (at 7am) after collection of the 48 hour PK sample. The subject will be instructed to return for the next treatment period or for the final follow-up visit, as appropriate. The final follow-up visit will occur 35 days after the last dose of study drug. Subjects will be assigned to each of the two treatments randomly as per the randomization schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests, 12 lead ECG and chest-x-ray. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Medical Investigator agrees that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with total T4 (4.5 -12.0 µg/dL), T3 (0.79 - 1.49 ng/mL) and TSH (21 weeks - 20 years: 0.7 - 6.4 µIU/mL, 21 - 54 years: 0.4 - 4.2 µIU/mL) values outside the normal range should always be excluded from enrollment (Interpath Lab Instructions, 2010).
2. Males between 18 and 50 years of age (both inclusive), who are willing to participate in the study and provide a written signed and dated informed consent.
3. Body weight more than or equal to 60 kg and BMI within the range 18.5-24.9 kg/m2 (inclusive).
4. Availability of a study volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.

Exclusion Criteria:

1. A positive pre-study urine drug screen.
2. A positive test for HIV antibody.
3. Subject has clinically significant abnormal values of laboratory parameters.
4. Regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
5. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
6. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
7. Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety.
8. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator contraindicates their participation.
9. Where participation in another study would result in donation of blood or blood products in excess of 350 ml within a 90 day period prior to this study.
10. Unwillingness or inability to follow the procedures outlined in the protocol.
11. Subject is mentally or legally incapacitated or the subject is incapable of understanding the informed consent.
12. Subject has any evidence of impaired renal, hepatic, cardiac, lung or gastrointestinal function. Study volunteers with a history of tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma will not be eligible for the study.
13. History of sensitivity to heparin or heparin-induced thrombocytopenia.
14. Regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
15. Subject is intolerant to venipuncture.
16. Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices] from 7 days prior to the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) and Area under concentration-time curve [AUC (0-48)] | -0.5, -0.25, 0, 0.5, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 18.00, 24.00 and 48.00 hours.
  Cmax and AUC (0-48) will be determined from the individual and mean serum concentration-time profiles of total T4 and T3, after adjustment by baseline levels of endogenous T4.

SECONDARY OUTCOMES:
Cmax | -0.5, -0.25, 0, 0.5, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 18.00, 24.00 and 48.00 hours.
  Cmax of serum T4 and T3 without adjustment by baseline levels of endogenous T4.
AUC (0-48) | -0.5, -0.25, 0, 0.5, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 18.00, 24.00 and 48.00 hours.
  AUC (0-48) of serum T4 and T3 without adjustment by baseline levels of endogenous T4.
Tmax | -0.5, -0.25, 0, 0.5, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 18.00, 24.00 and 48.00 hours.
  Tmax of serum T4 and T3 with and without adjustment by baseline levels of endogenous T4.
Kel | -0.5, -0.25, 0, 0.5, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 18.00, 24.00 and 48.00 hours.
  Kel of serum T4 and T3 with and without adjustment by baseline levels of endogenous T4.
t1/2 | -0.5, -0.25, 0, 0.5, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 18.00, 24.00 and 48.00 hours.
  t1/2 of serum T4 and T3 with and without adjustment by baseline levels of endogenous T4.
Serum TSH | At 12 hours pre-dose and 48 hours post dose
  Change in serum TSH
Adverse events | Up to 70 days after initiation of study
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hyderabad, India